CLINICAL TRIAL: NCT00049673
Title: A Randomized Phase III Study Of Thalidomide And Prednisone As Maintenance Therapy Following Autologous Stem Cell Transplant in Patients With Multiple Myeloma
Brief Title: Thalidomide and Prednisone After Autologous Stem Cell Transplantation Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MY10; CAN-NCIC-JMY10 (Other: PDQ); ECOG-NCIC-JMY10 (Other: ECOG); CELGENE-CAN-NCIC-MY10 (Other: Celgene); CDR0000258158 (Other: PDQ)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Prednisone; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Experimental): Patients receive oral thalidomide daily and oral prednisone every other day for 4 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: prednisone; Drug: thalidomide
- Arm II (No Intervention): Patients undergo observation.

INTERVENTIONS:
Drug: prednisone — Given orally
  Arms: Arm I
Drug: thalidomide — Given orally
  Arms: Arm I

SUMMARY:
RATIONALE: Thalidomide may stop the growth of multiple myeloma by stopping blood flow to the tumor. It is not yet known whether combining thalidomide with prednisone and giving them after autologous stem cell transplantation may be effective in treating multiple myeloma.

PURPOSE: This randomized phase III trial is studying thalidomide and prednisone to see how well they work compared to observation in treating patients who have undergone stem cell transplantation for multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare overall survival of patients with multiple myeloma treated with thalidomide and prednisone as maintenance therapy vs observation alone after autologous stem cell transplantation.
* Compare progression-free survival of patients treated with these regimens.
* Compare quality of life of patients treated with these regimens.
* Compare toxic effects of these regimens in these patients.
* Compare the objective venous thromboembolism rate in symptomatic patients treated with these regimens.

OUTLINE: This is a randomized, non-blinded, multicenter study. Patients are stratified according to treatment center, age (under 60 vs 60 and over), and response to prior transplantation (complete vs incomplete). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral thalidomide daily and oral prednisone every other day for 4 years in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo observation.

For both arms, patients are assessed (including for quality of life) regularly throughout the treatment/observation period: at baseline, every 2 months for 6 months, every 3 months for up to 4 years, and then annually thereafter.

After the treatment/observation period, patients are followed annually..

PROJECTED ACCRUAL: A total of 324 patients will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed multiple myeloma as evidenced by one of the following:

  * Biopsy of an osteolytic lesion or soft tissue tumor composed of plasma cells
  * Bone marrow aspirate and/or biopsy demonstrating at least 10% plasmacytosis
  * Bone marrow less than 10% plasma cells with at least 1 bony lesion and meets the M-protein criteria as below
* Detectable serum M-component of IgG, IgA, IgD, or IgE at initial diagnosis OR
* Urinary excretion of light chain (Bence Jones) protein at least 1.0 gm/24 hrs if only light chain disease (urine M-protein) was present at initial diagnosis
* Previously treated with autologous stem cell transplantation after high-dose melphalan (200 mg/m^2) within the past 60-100 days

  * Received transplantation within 1 year of the beginning of initial chemotherapy for multiple myeloma
  * No evidence of disease progression

PATIENT CHARACTERISTICS:

Age

* 16 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Hematopoietic

* No prior hereditary hypercoaguable disorder
* Granulocyte count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST and/or ALT no greater than 2 times ULN
* Alkaline phosphatase no greater than 2 times ULN

Renal

* Creatinine no greater than 3 times ULN

Cardiovascular

* No prior spontaneous deep vein thrombosis within the past 5 years

  * Catheter-associated thrombus allowed
* No uncontrolled hypertension

Pulmonary

* No prior pulmonary embolism within the past 5 years

Other

* No other prior or concurrent malignancy except adequately treated squamous cell or basal cell skin cancer or carcinoma in situ of the cervix or any cancer treated more than 5 years prior to study entry and presumed cured
* No prior gastric ulceration or bleeding within the past 5 years
* No prior documented lupus anti-coagulant or anti-phospholipid antibody
* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use 2 effective methods of contraception for 1 month prior, during, and 1 month after study participation
* Male patients must use effective barrier contraception during and for 1 month after study participation
* No avascular necrosis of the hips or shoulders
* No grade 2 or greater peripheral neuropathy causing symptomatic dysfunction (vincristine-induced sensory symptoms allowed)
* No diabetes with end-organ damage defined as:

  * Documented diabetic neuropathy
  * Retinal vascular proliferation requiring treatment
  * Cardiovascular disease requiring active therapy
* Willing to complete quality of life questionnaires
* Employment does not prohibit the use of sedatives
* No other major medical illness or condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior double autologous or allogeneic hematopoietic stem cell transplantation
* No prior thalidomide

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No other concurrent anti-cancer therapy
* No other concurrent investigational therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2002-10-15 (Actual); Primary Completion 2011-10-19 (Actual); Study Completion 2013-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Keith Stewart, MD, Study Chair — Mayo Clinic; Martha Q. Lacy, MD, Study Chair — Mayo Clinic
Locations (18):
- Canada (18):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - CHA-Hopital Du St-Sacrement, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stewart AK, Trudel S, Bahlis NJ, White D, Sabry W, Belch A, Reiman T, Roy J, Shustik C, Kovacs MJ, Rubinger M, Cantin G, Song K, Tompkins KA, Marcellus DC, Lacy MQ, Sussman J, Reece D, Brundage M, Harnett EL, Shepherd L, Chapman JA, Meyer RM. A randomized phase 3 trial of thalidomide and prednisone as maintenance therapy after ASCT in patients with MM with a quality-of-life assessment: the National Cancer Institute of Canada Clinicals Trials Group Myeloma 10 Trial. Blood. 2013 Feb 28;121(9):1517-23. doi: 10.1182/blood-2012-09-451872. Epub 2013 Jan 7. PMID 23297129
- [Derived] Kovacs MJ, Davies GA, Chapman JA, Bahlis N, Voralia M, Roy J, Kouroukis CT, Chen C, Belch A, Reece D, Zhu L, Meyer RM, Shepherd L, Stewart KA. Thalidomide-prednisone maintenance following autologous stem cell transplant for multiple myeloma: effect on thrombin generation and procoagulant markers in NCIC CTG MY.10. Br J Haematol. 2015 Feb;168(4):511-7. doi: 10.1111/bjh.13176. Epub 2014 Oct 10. PMID 25302852

RESULTS

PARTICIPANT FLOW:
Groups:
- Prednisone: Patients receive oral thalidomide daily and oral prednisone every other day for 4 years in the absence of disease progression or unacceptable toxicity.
  prednisone: Given orally
  thalidomide: Given orally
- Observation: Patients undergo observation.
Period: Overall Study
Arm/Group | Prednisone | Observation
Started | 166 | 166
Completed | 165 | 163
Not Completed | 1 | 3
Not completed — No receive treatment/lost to follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisone | Observation | Total
Number analyzed (Participants) | 166 | 166 | 332
Age, Customized [Count of Participants; unit: Participants]
  Age < 60 | 102 | 103 | 205
  Age > or = 60 | 64 | 63 | 127
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 56 | 114
  Male | 108 | 110 | 218
Region of Enrollment [Number; unit: participants]
  Canada | 162 | 162 | 324
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Number of patients died from any cause during the study.
Time Frame: 9 years
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisone | Observation
Number analyzed (Participants) | 166 | 166
Participants
  Death | 50 | 61
  Alive | 116 | 105
Statistical Analysis 1: Comparison: Prednisone vs Observation; Test type: Superiority; p = 0.18, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.53 to 1.14]

2. Secondary Outcome: Disease Progression-free Survival
Description: Number of patients with disease progression or death
Time Frame: 9 years
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisone | Observation
Number analyzed (Participants) | 166 | 166
Participants
  Disease progression | 100 | 127
  Without progression | 66 | 39
Statistical Analysis 1: Comparison: Prednisone vs Observation; Test type: Superiority; p = 0.0001, Log Rank; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.43 to 0.73]

ADVERSE EVENTS:
Time Frame: 9 years
Arm/Group | Prednisone | Observation
All-Cause Mortality (participants affected / at risk) | 50/165 | 61/163
Serious Adverse Events (participants affected / at risk) | 5/165 | 2/163
Other Adverse Events (participants affected / at risk) | 165/165 | 158/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prednisone (N=165) | Observation (N=163)
Sinus bradycardia (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Other (Immune system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prednisone (N=165) | Observation (N=163)
Edema (Cardiac disorders) | 72 | 29
Inner ear/hearing (Ear and labyrinth disorders) | 25 | 4
Cushingoid appearance (Endocrine disorders) | 25 | 0
Blurred vision (Eye disorders) | 31 | 5
Cataract (Eye disorders) | 18 | 1
Constipation (Gastrointestinal disorders) | 97 | 32
Diarrhea (Gastrointestinal disorders) | 31 | 36
Mouth dryness (Gastrointestinal disorders) | 55 | 5
Dyspepsia/heartburn (Gastrointestinal disorders) | 41 | 17
Nausea (Gastrointestinal disorders) | 37 | 28
Stomatitis (Gastrointestinal disorders) | 14 | 9
Vomiting (Gastrointestinal disorders) | 16 | 19
Other (Gastrointestinal disorders) | 23 | 6
Abdominal pain (Gastrointestinal disorders) | 30 | 24
Fatigue (General disorders) | 120 | 95
Other (General disorders) | 28 | 23
Chest pain (General disorders) | 18 | 7
Pain-Other (General disorders) | 45 | 22
Allergic reaction (Immune system disorders) | 12 | 6
Fever (Immune system disorders) | 22 | 16
Other (Immune system disorders) | 20 | 11
Infection w/o neutropen (Infections and infestations) | 113 | 88
Infection-unknown ANC (Infections and infestations) | 11 | 7
Bruising (Injury, poisoning and procedural complications) | 14 | 1
Hypercholesterolemia (Investigations) | 15 | 3
Anorexia (Metabolism and nutrition disorders) | 16 | 15
Muscle weakness (Musculoskeletal and connective tissue disorders) | 32 | 9
Other (Musculoskeletal and connective tissue disorders) | 34 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 40
Myalgia (Musculoskeletal and connective tissue disorders) | 74 | 51
Bone pain (Musculoskeletal and connective tissue disorders) | 119 | 121
Taste disturbance (Nervous system disorders) | 15 | 7
Dizziness (Nervous system disorders) | 70 | 15
Memory loss (Nervous system disorders) | 19 | 3
Neuropathy-motor (Nervous system disorders) | 13 | 4
Neuropathy-sensory (Nervous system disorders) | 147 | 71
Depressed conscious. (Nervous system disorders) | 29 | 5
Tremor (Nervous system disorders) | 33 | 2
Headache (Nervous system disorders) | 24 | 19
Neuropathic pain (Nervous system disorders) | 16 | 12
Anxiety (Psychiatric disorders) | 63 | 22
Confusion (Psychiatric disorders) | 17 | 2
Insomnia (Psychiatric disorders) | 69 | 44
Depression (Psychiatric disorders) | 28 | 27
Urine frequency/urgency (Renal and urinary disorders) | 14 | 12
Erectile impotence (Reproductive system and breast disorders) | 11 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 38
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 69 | 33
Other (Respiratory, thoracic and mediastinal disorders) | 13 | 7
Sweating (Skin and subcutaneous tissue disorders) | 27 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 28 | 17
Nail changes (Skin and subcutaneous tissue disorders) | 9 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 16
Rash/desquamation (Skin and subcutaneous tissue disorders) | 60 | 39
Other (Skin and subcutaneous tissue disorders) | 14 | 11
Hypertension (Vascular disorders) | 27 | 13
Thrombosis/embolism (Vascular disorders) | 12 | 1
Hot flashes/ flushes (Vascular disorders) | 15 | 6
Flushing (Vascular disorders) | 9 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No